CLINICAL TRIAL: NCT01847885
Title: A Randomized, Double-Blinded, Placebo-Control Multicenter Pivotal Study of the Smartpatch Peripheral Nerve Stimulation (PNS) System for the Treatment of Chronic Post-Stroke Shoulder Pain
Brief Title: Electrical Stimulation for the Treatment of Chronic Post-Stroke Shoulder Pain Using the Smartpatch System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0131-CSP-000
Record Dates: First submitted 2013-04-23; First posted 2013-05-07 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Post-stroke Shoulder Pain; Hemiplegic Shoulder Pain
Keywords: electrical stimulation; neurostimulation; neuromodulation; post-stroke shoulder pain; hemiplegic shoulder pain
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smartpatch Treatment Group (Experimental): Subjects in the Treatment Group will have a Smartpatch Lead placed in the shoulder, will use the Smartpatch Peripheral Nerve Stimulation (PNS) System, and will receive electrical stimulation.
  Interventions: Device: Smartpatch Peripheral Nerve Stimulation (PNS) System
- Smartpatch Control Group (Sham Comparator): Subjects in the Control Group will have a Smartpatch Lead placed in the shoulder, will use the Smartpatch Peripheral Nerve Stimulation (PNS) System, but will not receive any electrical stimulation.
  Interventions: Device: Smartpatch Peripheral Nerve Stimulation (PNS) System

INTERVENTIONS:
Device: Smartpatch Peripheral Nerve Stimulation (PNS) System — The Smartpatch System is an Investigation Device which delivers mild electrical stimulation to the muscles in the shoulder. The Smartpatch System includes a small wire (called a "Lead") that is placed through the skin into the muscle of the shoulder. It also includes a device worn on the body that delivers stimulation (called the Smartpatch Stimulator).
  Other Names: Smartpatch System, Smartpatch

SUMMARY:
The purpose of this study is to determine if electrical stimulation (small levels of electricity) reduces post-stroke shoulder pain. This study involves a device called the Smartpatch System. The Smartpatch System delivers mild electrical stimulation to the muscles in the shoulder. The Smartpatch System includes a small wire (called a "Lead") that is placed through the skin into the muscle of the shoulder. It also includes a device worn on the body that delivers stimulation (called the Smartpatch Stimulator).

ELIGIBILITY:
Key Inclusion Criteria:

* At least 21 years of age
* Post-stroke shoulder pain
* At least 6 months after stroke that caused shoulder pain

Key Exclusion Criteria:

* Use of habit-forming (narcotic) medications
* Bleeding disorder
* History of recurrent skin infections
* Parkinson's Disease, Spinal Cord Injury, traumatic brain injury, Multiple Sclerosis, or Complex Regional Pain Syndrome
* Heart arrhythmia or artificial heart valves
* Uncontrolled seizures
* Implanted Electronic Device
* Pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08-21 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Kessler Foundation Research Center, West Orange, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - Carolinas Rehabilitation/Carolinas Healthcare, Charlotte, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in March 2013 and was concluded in May 2015. Subjects were screened for the study from the available pool of candidates who presented to the Investigators with shoulder pain following stroke.
Pre-assignment Details: Following informed consent and enrollment in the study, subjects were given a 7-day diary to complete at home. At the following visit, subjects were randomized once all eligibility criteria were met. Therefore it was possible for subjects to no longer meet eligibility criteria or drop out after enrollment, but prior to being randomized.
Groups:
- Enrolled Subjects: Subjects who signed a consent form.
- Smartpatch Treatment Group (Full Analysis Set): Subjects in the Treatment Group had a Smartpatch Lead placed in the shoulder, used the Smartpatch Peripheral Nerve Stimulation (PNS) System, and received electrical stimulation.
- Smartpatch Control Group (Full Analysis Set): Subjects in the Control Group had a Smartpatch Lead placed in the shoulder, used the Smartpatch Peripheral Nerve Stimulation (PNS) System, but did not receive any electrical stimulation.
Period: Initial Enrollment (Consented)
Arm/Group | Enrolled Subjects | Smartpatch Treatment Group (Full Analysis Set) | Smartpatch Control Group (Full Analysis Set)
Started | 88 | 0 | 0
Randomized (Subjects who signed a consent form, met all eligibility criteria, and were randomized.) | 46 | 0 | 0
Full Analysis Set (Subjects who were consented, randomized, and met all eligibility criteria prior to lead placement) | 43 | 0 | 0
Safety Set (Subjects who received a Lead.) | 41 | 0 | 0
Per Protocol Set (Subjects who received a Lead, had enough scores in the diary, and met eligibility through treatment.) | 40 | 0 | 0
Completed | 40 | 0 | 0
Not Completed | 48 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Screen failure | 39 | 0 | 0
Not completed — Pending prior to enrollment stop | 6 | 0 | 0
Period: Randomization
Arm/Group | Enrolled Subjects | Smartpatch Treatment Group (Full Analysis Set) | Smartpatch Control Group (Full Analysis Set)
Started | 0 | 31 | 15
Full Analysis Set | 0 | 28 | 15
Safety Set | 0 | 28 | 13
Per Protocol Set | 0 | 27 | 13
Completed | 0 | 27 | 13
Not Completed | 0 | 4 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Screen Failure | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set includes all randomized patients who continued to meet all eligibility criteria prior to the time of lead placement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Smartpatch Treatment Group (Full Analysis Set) | Smartpatch Control Group (Full Analysis Set) | Total
Number analyzed (Participants) | 28 | 15 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (11.8) | 58.9 (9.8) | 57.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 18 | 9 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 25 | 15 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 1 | 11
  White | 15 | 11 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Type of stroke [Count of Participants; unit: Participants] — Medical type of stroke, either hemorrhagic or ischemic
  Participants
    Hemorrhagic | 11 | 5 | 16
    Ischemic | 16 | 10 | 26
    Unknown/not collected | 1 | 0 | 1
Time elapsed from stroke, years [Mean (Standard Deviation); unit: years] — Years elapsed from the date of stroke to enrollment in the study
  years | 5.1 (4.7) | 3.5 (2.8) | 4.5 (4.2)
Presence of shoulder subluxation [Count of Participants; unit: Participants] — Population: Subjects were evaluated to determine the presence or absence of shoulder subluxation (partial or incomplete dislocation of shoulder). Of note, this analysis is on the safety set (subjects who received a Smartpatch lead where n=41).
  Participants
    Subluxation present: number analyzed (Participants) | 28 | 13 | 41
    Subluxation present | 23 | 11 | 34
    Subluxation absent: number analyzed (Participants) | 28 | 13 | 41
    Subluxation absent | 5 | 2 | 7
Beck Depression Inventory score [Mean (Standard Deviation); unit: Beck Depression Score] — The Beck Depression Inventory, version II is a survey used to measure depression severity. Scores from 0-13 indicate minimal depression, 14-19 mild depression, 20-28 moderate depression, and 29-63 severe depression. The score range is 0 to 63.
  Beck Depression Score | 13.2 (9.0) | 17.6 (11.9) | 14.7 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Shoulder Pain Intensity at End of Treatment (EOT)
Description: A diary was used in the study to capture daily worst shoulder pain intensity over a 7-day period. The diary included a pain intensity question asked each day to the subject. The pain intensity question is excerpted from the Brief Pain Inventory - Short Form Question 3 (BPI-3) and is stated as "please rate your pain by circling the one number that best describes your pain at its worst in the last 24 hours". BPI-3 is a scale of 0 to 10 where 0 represents no pain and 10 represents worst pain. The median scores were calculated for each diary period. The median diary score at End of Treatment (EOT) was compared to the median baseline diary score to calculate the change in pain intensity. The group mean of the median scores for treatment was compared to the group mean of the medians scores for the control group at baseline and at EOT.
Time Frame: Baseline, End of Treatment (4-weeks of Treatment/Control)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Smartpatch Treatment Group (Full Analysis Set) | Smartpatch Control Group (Full Analysis Set)
Number analyzed (Participants) | 28 | 15
scores on a scale
  Baseline diary score | 7.1 (1.5) | 6.6 (1.5)
  EOT diary score | 4.1 (2.3) | 4.1 (3.1)
  Change in pain intensity from baseline | 3.1 (2.3) | 2.5 (3.1)

2. Primary Outcome: Number of Participants With Device Related Adverse Event Rates in Treatment and Control Groups
Description: At each study visit following the baseline assessment, subjects were questioned if any changes in their medical status or condition had occurred. If the change was an adverse event, an adverse event form was completed by the site.
Time Frame: 16 weeks total - 4 weeks from baseline visit to EOT visit, followed by 12 weeks post-treatment
Population: Safety set
Measure: Number; unit: device related adverse events
Groups:
- Smartpatch Treatment Group (Safety Set): Subjects in the Treatment Group had a Smartpatch Lead placed in the shoulder, used the Smartpatch Peripheral Nerve Stimulation (PNS) System, and received electrical stimulation.
- Smartpatch Control Group (Safety Set): Subjects in the Control Group had a Smartpatch Lead placed in the shoulder, used the Smartpatch Peripheral Nerve Stimulation (PNS) System, but did not receive any electrical stimulation.
Arm/Group | Smartpatch Treatment Group (Safety Set) | Smartpatch Control Group (Safety Set)
Number analyzed (Participants) | 28 | 13
device related adverse events | 16 | 3

3. Secondary Outcome: Change From Baseline Shoulder Pain Interference at End of Treatment
Description: The degree to which shoulder pain interferes with daily activities was assessed using Question 9 of the Brief Pain Inventory (BPI-9) collected from the BPI Short Form administered during clinic visits. This question asks the subject to rate the degree to which their pain has interfered with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life on a scale of 0 to 10, where 0 is "does not interfere" and 10 is "completely interferes" within the last week. The mean of these seven scores will be calculated to obtain the pain interference score.
Time Frame: Baseline, End of Treatment (4-weeks of Treatment/Control)
Population: Per protocol set (Subjects in the full analysis set who also were implanted with a Smartpatch Lead, had an adequate number of worst pain intensity (BPI3) scores in the End of Treatment subject diary period, and continued to meet all eligibility criteria throughout treatment).
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Smartpatch Treatment Group (Per Protocol Set): Subjects in the Treatment Group had a Smartpatch Lead placed in the shoulder, used the Smartpatch Peripheral Nerve Stimulation (PNS) System, and received electrical stimulation.
- Smartpatch Control Group (Per Protocol Set): Subjects in the Control Group had a Smartpatch Lead placed in the shoulder, used the Smartpatch Peripheral Nerve Stimulation (PNS) System, but did not receive any electrical stimulation.
Arm/Group | Smartpatch Treatment Group (Per Protocol Set) | Smartpatch Control Group (Per Protocol Set)
Number analyzed (Participants) | 27 | 13
scores on a scale
  Baseline score | 4.8 (2.4) | 5.0 (2.0)
  EOT score | 1.8 (1.8) | 2.6 (3.3)
  Change in pain interference from baseline | 3.1 (2.2) | 2.4 (2.7)

4. Secondary Outcome: Durability of Change From Baseline Shoulder Pain Intensity at 12-weeks Beyond Treatment
Description: A diary was used in the study to capture daily worst shoulder pain intensity over a 7-day period. The diary included a pain intensity question asked each day to the subject. The pain intensity question is excerpted from the Brief Pain Inventory - Short Form Question 3 (BPI-3) and is stated as "please rate your pain by circling the one number that best describes your pain at its worst in the last 24 hours". BPI-3 is a scale of 0 to 10 where 0 represents no pain and 10 represents worst pain. The median scores were calculated for each diary period. The median diary score at 12 weeks post-treatment was compared to the median baseline diary score to calculate the change in pain intensity. The group mean of the median scores for 12 weeks post-treatment was compared to the group mean of the median scores for the control group at baseline.
Time Frame: Baseline, 12-wks post-treatment
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Smartpatch Treatment Group (Full Analysis Set) | Smartpatch Control Group (Full Analysis Set)
Number analyzed (Participants) | 28 | 15
scores on a scale
  Baseline diary score | 7.1 (1.5) | 6.6 (1.5)
  12- weeks post-treatment diary score | 4.3 (2.9) | 4.3 (2.5)

5. Secondary Outcome: Change From Baseline Quality of Life at End of Treatment
Description: The Medical Outcomes Study Short Form (SF-36v2) was administered at clinic visits to assess the impact of peripheral nerve stimulation on the subject's health-related quality of life. The SF-36v2 is a generic health survey designed to assess basic physical functioning and emotional well-being regardless of the disease or treatment. The 36 questions were grouped into two components: physical and mental. The survey was scored using norm-based scoring algorithm where a score of 0 indicates maximum disability and a score of 100 indicates no disability. Change in each component score was derived from End of Treatment score minus baseline score.
Time Frame: Baseline, End of Treatment (4-weeks of Treatment/Control)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Smartpatch Treatment Group (Per Protocol Set) | Smartpatch Control Group (Per Protocol Set)
Number analyzed (Participants) | 27 | 13
scores on a scale
  Physical Component Baseline score | 38.0 (8.9) | 35.4 (10.4)
  Change in Physical Component score from baseline | 4.8 (7.0) | 3.5 (9.3)
  Mental Component Baseline score | 54.3 (10.7) | 47.9 (9.5)
  Change in Mental Component score from baseline | 4.1 (10.1) | 9.1 (13.2)

6. Secondary Outcome: Change From Baseline Average Pain Intensity at End of Treatment
Description: A diary was used in the study to capture daily average shoulder pain intensity over a 7-day period. The diary included a pain intensity question asked each day to the subject. The pain intensity question is excerpted from the Brief Pain Inventory - Short Form Question 5 (BPI-5) and is stated as "please rate your pain by circling the one number that best describes your pain on the average". BPI-5 is a scale of 0 to 10 where 0 represents no pain and 10 represents worst pain. The mean scores were calculated for each diary period. The mean diary score at End of Treatment (EOT) was compared to the mean baseline diary score to calculate the change in pain intensity.
Time Frame: Baseline, End of Treatment (4-weeks of Treatment/Control)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Smartpatch Treatment Group (Per Protocol Set) | Smartpatch Control Group (Per Protocol Set)
Number analyzed (Participants) | 27 | 13
scores on a scale
  Baseline diary score | 5.2 (2.0) | 4.8 (1.7)
  EOT diary score | 2.6 (1.8) | 2.4 (2.2)
  Change in pain intensity from baseline | 2.7 (2.3) | 2.5 (2.3)

7. Secondary Outcome: Patient Global Impression of Change at End of Treatment
Description: The Patient Global Impression of Change (PGIC) scale was administered at EOT to assess subject perception of overall improvement and patient preferences. The PGIC scale asks subjects to rate their improvement with treatment on a 7-point scale (centered at 4) that ranges from "very much worse" to "very much improved" relative to baseline.
Time Frame: End of Treatment (4-weeks of Treatment/Control)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Smartpatch Treatment Group (Per Protocol Set) | Smartpatch Control Group (Per Protocol Set)
Number analyzed (Participants) | 27 | 13
Participants
  Very much worse | 0 | 0
  Much worse | 0 | 0
  Minimally worse | 0 | 2
  No change | 1 | 2
  Minimally improved | 11 | 5
  Much improved | 13 | 3
  Very much improved | 2 | 1

8. Secondary Outcome: Change in Pain Medication Usage at End of Treatment
Description: Subjects completed 7-day diaries, in which they listed all pain medications they took during the 7 days. A blinded third party medication committee reviewed medications collected for each 7-day diary period and scored medication changes, in comparison to the baseline diary medications as "no change" (no change in dosage or change is not clinically meaningful to impact pain outcomes), "increase" (clinically meaningful increase in medication that would impact pain outcomes), or "decrease" (clinically meaningful decrease in medication that would impact pain outcomes).
Time Frame: End of Treatment (4-weeks of Treatment/Control)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Smartpatch Treatment Group (Per Protocol Set) | Smartpatch Control Group (Per Protocol Set)
Number analyzed (Participants) | 25 | 13
Participants
  Decrease in pain med usage compared to baseline | 6 | 4
  No change in pain med usage compared to baseline | 16 | 8
  Increase in pain med usage compared to baseline | 3 | 1

9. Secondary Outcome: Clinical Global Impression of Improvement at End of Treatment
Description: The Blinded Evaluator rated each subject enrolled at their site using a question adapted from the Clinical Global Impression (CGI) scale, known as the Clinical Global Impression-Improvement scale (CGI-I). For the CGI-I, a Blinded Evaluator was asked to rate the subject's total improvement compared to their condition at baseline. The CGI-I uses a 7-point scale (centered at 4) that ranges from "very much worse" to "very much improved".
Time Frame: End of Treatment (4-weeks of Treatment/Control)
Population: Per protocol set (Subjects in the full analysis set who also were implanted with a Smartpatch Lead, had an adequate number of worst pain intensity (BPI3) scores in the End of Treatment subject diary period, and continued to meet all eligibility criteria throughout treatment). The CGI-I was not completed for one subject in the treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Smartpatch Treatment Group (Per Protocol Set) | Smartpatch Control Group (Per Protocol Set)
Number analyzed (Participants) | 26 | 13
Participants
  Very much worse | 0 | 0
  Much worse | 0 | 0
  Minimally worse | 0 | 1
  No change | 1 | 3
  Minimally improved | 11 | 4
  Much improved | 10 | 5
  Very much improved | 4 | 0

10. Other Pre Specified Outcome: User Satisfaction With The Smartpatch System at End of Treatment
Description: Subjects completed the sponsor-developed Subject Satisfaction Survey at the End of Treatment (EOT) visit. The results of these surveys demonstrate the usability of the Smartpatch System and subject satisfaction with treatment.
Time Frame: End of Treatment (4-weeks of Treatment/Control)
Population: Safety set (Subjects who were implanted with a Smartpatch Lead)
Measure: Count of Participants; unit: Participants
Arm/Group | Smartpatch Treatment Group (Safety Set) | Smartpatch Control Group (Safety Set)
Number analyzed (Participants) | 28 | 13
Participants
  Reported study had positive impact on their life | 27 | 9
  Reported being satisfied with experience in study: number analyzed (Participants) | 28 | 12
  Reported being satisfied with experience in study | 27 | 10
  Would recommend participation in study to a friend: number analyzed (Participants) | 28 | 11
  Would recommend participation in study to a friend | 28 | 11
  Tolerated lead placement with no discomfort | 16 | 8
  Tolerated lead placement with some discomfort | 11 | 5
  Tolerated lead placement with a lot of discomfort | 1 | 0

11. Other Pre Specified Outcome: User Satisfaction With The Smartpatch System at 12-weeks Beyond Treatment
Description: Subjects completed the sponsor-developed Subject Satisfaction Survey at the end of the 12-week post-treatment period. The results of these surveys demonstrate the usability of the Smartpatch System and subject satisfaction with treatment.
Time Frame: 12-week post-treatment
Population: Safety set (Subjects who were implanted with a Smartpatch Lead)
Measure: Count of Participants; unit: Participants
Arm/Group | Smartpatch Treatment Group (Safety Set) | Smartpatch Control Group (Safety Set)
Number analyzed (Participants) | 28 | 13
Participants
  Reported study had positive impact on their life | 27 | 11
  Reported being satisfied with experience in study | 26 | 11
  Would recommend participation in study to a friend | 28 | 13
  Tolerated lead placement with no discomfort | 20 | 9
  Tolerated lead placement with some discomfort | 7 | 4
  Tolerated lead placement with a lot of discomfort | 1 | 0

12. Other Pre Specified Outcome: Performance of the Smartpatch System
Description: A sponsor-developed Clinician Satisfaction Survey was administered to the Investigator(s) at each site performing lead placement and included questions pertaining to use of the Smartpatch device as well as the overall impression of the therapy.
Time Frame: At completion of study, approximately 2.5 years
Population: "Count of participants" represents Investigators responding to the survey rather than study participants.
Measure: Count of Participants; unit: Participants
Groups:
- Investigators: Investigator(s) at each site performing lead placement
Arm/Group | Investigators
Number analyzed (Participants) | 7
Participants
  Agreed time to perform procedure was acceptable | 7
  Agreed that device components performed well | 6
  Agreed that patients tolerated the procedure well | 6
  Agreed that the Smartpatch System was easy to use | 7
  Liked the size, weight, & shape of the Stimulator | 7
  Agreed study beneficial for most of their patients | 5

13. Post Hoc Outcome: Composite 30% Reduction in Pain Intensity or Pain Interference From Baseline to End of Treatment (EOT)
Description: Subjects who reported an reduction of at least 30% in either pain intensity or pain interference from baseline to End of Treatment (EOT) using the Brief Pain Inventory (BPI) Short Form.
  The pain intensity score is excerpted from BPI question 3, worst pain, taken from 7-day diaries. This scale ranges from 0 representing no pain to 10 representing worst pain. The median diary score at EOT was compared to the median baseline diary score to calculate the percentage of subjects who had at least a 30% reduction in pain intensity.
  Pain interference was assessed using BPI question 9. Subjects rated the degree to which their pain interfered with seven facets of daily life on a scale of 0 to 10, where 0 is "does not interfere" and 10 is "completely interferes". The mean of these 7 scores was calculated to obtain the pain interference score. The score at EOT was compared to the baseline score to determine the percentage of subjects who had at least a 30% reduction in pain interference.
Time Frame: 4 weeks (from baseline visit to EOT visit)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Smartpatch Treatment Group (Per Protocol Set) | Smartpatch Control Group (Per Protocol Set)
Number analyzed (Participants) | 27 | 13
Participants | 25 | 8

14. Post Hoc Outcome: 30% Reduction in Pain Interference From Baseline to End of Treatment (EOT)
Description: The degree to which shoulder pain interferes with daily activities was assessed using Question 9 of the Brief Pain Inventory (BPI-9) collected from the BPI Short Form administered during clinic visits. This question asks the subject to rate the degree to which their pain has interfered with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life on a scale of 0 to 10, where 0 is "does not interfere" and 10 is "completely interferes" within the last week. The mean of these seven scores was calculated to obtain the pain interference score. The score at End of Treatment (EOT) was compared to the baseline score to determine the percentage of subjects who had a clinically significant (30% or greater) reduction in pain interference.
Time Frame: 4 weeks (from baseline visit to EOT visit)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Smartpatch Treatment Group (Per Protocol Set) | Smartpatch Control Group (Per Protocol Set)
Number analyzed (Participants) | 27 | 13
Participants | 24 | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 29 months (time from when the first subject was enrolled in April 2013 to when the last subject was completed in August 2015).
Description: At each study visit following the baseline assessment, subjects were questioned if any changes in their medical status or condition had occurred. If the change was an adverse event, an adverse event form was completed by the site.
Groups:
- Enrolled Subjects Who Did Not Receive the Study Device: Subjects who were consented, but were not randomized and did not receive the study device or any intervention.
Arm/Group | Enrolled Subjects Who Did Not Receive the Study Device | Smartpatch Treatment Group (Safety Set) | Smartpatch Control Group (Safety Set)
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/28 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/88 | 0/28 | 0/13
Other Adverse Events (participants affected / at risk) | 0/88 | 22/28 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects Who Did Not Receive the Study Device (N=88) | Smartpatch Treatment Group (Safety Set) (N=28) | Smartpatch Control Group (Safety Set) (N=13)
Focal seizure (occurred prior to receiving any intervention) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects Who Did Not Receive the Study Device (N=88) | Smartpatch Treatment Group (Safety Set) (N=28) | Smartpatch Control Group (Safety Set) (N=13)
General malaise after procedure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lead barb retained (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Mild bruising under lead connector (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Mild erythema or irritation at lead exit site (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Papule, lead exit site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation/dermatitis from bandages (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (12) | 4 (4)
Skin irritation/redness/or mild skin tears from Smartpatch Pad (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Double pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3)
New numbness to left lower extremity (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Lasik eye surgery (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Depression and suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Increased pain (in paretic shoulder, lower back, and left lower extremity) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness and headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study included a pre-planned interim analysis for sample size re-estimation. The study was suspended because the treatment effect (both groups experienced clinically significant reductions in pain) required a sample size more than 90 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less